CLINICAL TRIAL: NCT01694095
Title: Characterization of Geographic Atrophy Progression in Patients With Age-related Macular Degeneration
Brief Title: Evolution and Risk Factors Associated With Geographic Atrophy Progression
Acronym: GAIN
Status: Completed | Type: Observational
Sponsor: Institut de la Macula y la Retina (Other)
Responsible Party: Principal Investigator, Jordi Mones, MD, PhD, Institut de la Macula y la Retina
Other Study IDs: GAIN-002-10-2010
Record Dates: First submitted 2012-09-22; First posted 2012-09-26 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Geographic Atrophy
Keywords: Geographic atrophy, prognosis, risk factors, natural history
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with geographic atrophy

SUMMARY:
Age-related macular degeneration is one of the leading causes of blindness worldwide. The factors that induce the progression of geographic atrophy, the advanced form of dry age-related macular degeneration, remain poorly understood. The aims of this study are to describe the natural history of geographic atrophy and identify potential risk factors associated with a faster spread of atrophy that may be used to develop rational therapies.

DETAILED DESCRIPTION:
Age-related macular degeneration is the leading cause of blindness in developed countries. Geographic atrophy is the advanced form of dry age-related macular degeneration, and currently has no effective therapy. Little is known about the risk factors that drive the progression of geographic atrophy, and yet they are crucial to understand the mechanisms of the disease. Therefore, the identification of risk factors associated with a faster spread of atrophy may help contribute to identify the causes of the disease and, ultimately, to develop new therapeutic strategies to manage the disorder.

The current prospective, observational, natural history study has the following objectives:

* Describe the natural history of geographic atrophy in anatomic and visual terms
* Identify risk factors associated with a faster enlargement of atrophy

The main hypothesis is that lipofuscin accumulation at the borders of atrophy as seen with fundus autofluorescence imaging is associated with a faster progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* 50 years of age or older
* Uni or bilateral areas of geographic atrophy in the macula (as defined as areas devoid of retinal pigment epithelium measuring at least 0.5 disk areas on a 35º fundus photograph centered on field 2) secondary to age-related macular degeneration
* Willing to provide Informed consent

Exclusion Criteria:

* Other causes of geographic atrophy aside from age-related macular degeneration (ie, drug induced, central serous chorioretinopathy)
* Prior history of wet age-related macular degeneration
* Other significant concomitant macular diseases (ie, significant epiretinal membrane, stage II-IV macular hole)
* Previous treatment with macular laser photocoagulation, photodynamic therapy, antiangiogenic drugs or other treatments for wet age-related macular degeneration
* Intraocular surgery aside from phacoemulsification
* Inability to measure the full extent of the area of atrophy on a 35º fundus autofluorescence image centered on field 2
* Areas of geographic atrophy in direct contact with peripapillary areas of atrophy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with geographic atrophy
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2009-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Median/mean change in area of geographic atrophy as measured in mm2 with fundus autofluorescence on a 30º image centered on field 2 | From baseline to last follow-up
  For measures related to change in the area of atrophy, a multivariable model will be fit and will include as an independent variable (amongst other presumed risk factors) fundus autofluorescence patterns

SECONDARY OUTCOMES:
Median change in area of geographic atrophy as measured in square root of mm2 with fundus autofluorescence on a 30º image centered on field 2 | From baseline to last follow-up
  Exploratory analysis, either in the main publication or in another paper

OTHER OUTCOMES:
Median/mean change in best-corrected visual acuity as measured with an Early Treatment Diabetic Retinopathy Study chart | From baseline to last follow-up
Percentage of eyes developing new choroidal neovascularization in the study eye as evaluated with fluorescein angiography and spectral-domain optical coherence tomography | From baseline to last follow-up
Median/mean change in area of geographic atrophy as measured in mm2 with fundus autofluorescence on a 30º image centered on field 2 | From baseline to last follow-up
  Principal component analysis will be used to reduce the number of independent variables to increase, if possible, the power of the study to detect an association

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Monés, MD, PhD, Principal Investigator — Institut de la màcula i de la retina
Locations (1):
- Institut de la màcula i de la retina, Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Biarnes M, Mones J, Trindade F, Alonso J, Arias L. Intra and interobserver agreement in the classification of fundus autofluorescence patterns in geographic atrophy secondary to age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 2012 Apr;250(4):485-90. doi: 10.1007/s00417-011-1846-y. Epub 2011 Oct 28. PMID 22033626
- [Result] Mones J, Biarnes M, Trindade F. Hyporeflective wedge-shaped band in geographic atrophy secondary to age-related macular degeneration: an underreported finding. Ophthalmology. 2012 Jul;119(7):1412-9. doi: 10.1016/j.ophtha.2012.01.026. Epub 2012 Mar 21. PMID 22440276
- [Result] Mones J, Biarnes M, Trindade F, Arias L, Alonso J. Optical coherence tomography assessment of apparent foveal swelling in patients with foveal sparing secondary to geographic atrophy. Ophthalmology. 2013 Apr;120(4):829-36. doi: 10.1016/j.ophtha.2012.09.054. Epub 2013 Jan 3. PMID 23290986
- [Result] Biarnes M, Forero CG, Arias L, Alonso J, Mones J. Reappraisal of geographic atrophy patterns seen on fundus autofluorescence using a latent class analysis approach. Invest Ophthalmol Vis Sci. 2014 Nov 18;55(12):8302-8. doi: 10.1167/iovs.13-13542. PMID 25406275